CLINICAL TRIAL: NCT05315180
Title: A Phase 1，Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of BPI-421286 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1，Open-label Study of BPI-421286 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661311
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Malignant Neoplasms; Metastatic Cancer
Keywords: Antineoplastic Agents; KRAS; NSCLC; Colorectal Cancer; Pancreatic Cancer; KRAS G12C
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dose exploration (Experimental): Enrollment into the dose exploration cohorts may be from any eligible solid tumor type. Dose escalation will begin with 1-6 subjects treated at the lowest planned dose level. If no DLT is observed, dose escalation will continue to the next planned dose cohort
  Interventions: Drug: BPI-421286
- dose expansion (Experimental): dose expansion may proceed with 2 groups consisting of subjects with KRAS p.G12C mutant advanced solid tumors. Dose expansion in these 2 groups may be done concurrently
  Interventions: Drug: BPI-421286

INTERVENTIONS:
Drug: BPI-421286 — Characterize the pharmacokinetics (PK)，safety，effcicay of BPI-421286 following administration as an oral Tablet formulation

SUMMARY:
Evaluate the safety and tolerability of BPI-421286 in adult subjects with advanced solid tumors.

Estimate the maximum tolerated dose (MTD) and/or a recommended phase 2 dose (RP2D) in adult subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented, locally-advanced or metastatic malignancy
* Standard treatment is not available or patient declines
* Adequate organ function

Exclusion Criteria:

* Active brain metastases from non-brain tumors.
* Gastrointestinal (GI) tract disease causing the inability to take oral medication.
* Other protocol specified criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety and tolerability of BPI-421286 in subjects with advanced solid tumor malignancies | 20 months
  Number of subjects with treatment related adverse events
determine the recommended Phase II dose (RP2D) and preliminarily to develop a suitable dosing regimen | 20 months
  Number of subjects with dose limiting toxicity

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of BPI-421286 | 20 months
  Blood plasma concentration
To determine overall response rate (ORR),calculated as the proportion of subjects with confirmed complete (CR) or partial response (PR) to BPI-421286 | 20 months
  Evaluate clinical activity/efficacy of BPI-421286
To evaluate the duration of response (DOR) in subjects with CR or PR as best response | 20 months
  Evaluate clinical activity/efficacy of BPI-421286
to evaluate the disease control rate (DCR) | 20 months
  Evaluate clinical activity/efficacy of BPI-421286
To evaluate progression-free survival (PFS) following initiation of BPI-421286 | 20 months
  Evaluate clinical activity/efficacy of BPI-421286
To evaluate overall (OS) following initiation of BPI-421286 | 20 months
  Evaluate clinical activity/efficacy of BPI-421286

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Shun Lu, Ph.D, Shanghai, Shanghai Municipality
  - Dingzhi Huang, Ph.D, Tianjin, Tianjin Municipality
  - Wen Li, Ph.D, Hangzhou, Zhejiang
  - Yun Fan,Ph.D, Hangzhou, Zhejiang
  - Shun Lu, Ph.D, Shanghai

IPD SHARING:
Plan to Share IPD: No